CLINICAL TRIAL: NCT02478944
Title: Esophageal Motility Disease Screening in Patient With Suspicion or Diagnosis of IBD
Acronym: EMSIBD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Francesco Vitali, MD, University Hospital Erlangen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Gastrolabor-IBD UKE
Record Dates: First submitted 2014-11-05; First posted 2015-06-23 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory bowel disease; Manometry
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Manometry

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Inflammatory bowel disease (Experimental): Patients with Crohn's disease and ulcerative colitis undergoing manometry
  Interventions: Device: Manometry

INTERVENTIONS:
Device: Manometry — Flexible tube catheter pressure measurement of oesophageal contractions. Measurement without any sedation, transnasal

SUMMARY:
Aims: Prospective evaluation of patients with a suspicion or diagnosis of Inflammatory bowel disease (IBD) to evaluate osophageal motility before and during therapy

Material and methods: The investigators prospectively perform manometry in patients with or with symptoms consistent with IBD. The investigators evaluate esophageal motility with high resolution manometry before, during and after IBD therapy. Clinical data are also collected to find possible correlations. The study do not modify the planned IBD therapy, but observe motility findings.

DETAILED DESCRIPTION:
Oesophageal motility is measured with the high resolution manometry in order to detect pathologic peristaltic amplitude values among patient before and after therapy (mesalazine, steroids, biologicals) compared to the standard values detected among the normal population. Diagnosic intervention like oesophagoduodenoscopy, colonoscopy and stenosis ballon dilation are allowed as are part of the IBD therapy and follow up.

No other interventions are administered to participants during this study.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory bowel disease
* Suspicion of inflammatory bowel disease

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-12 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Manometry finding (peristaltic amplitude values mmHG) compared to normal population findings | 1 year
Correlation with gastrointestinal symptoms to manometry findings (peristaltic amplitude values) | 1 year

SECONDARY OUTCOMES:
Manometry findings (peristaltic amplitude values, mmHG) during therapy | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Albrecht, MD, Study Director — UK Erlangen
Locations (1):
- University Hospital Erlangen Nuremberg, Erlangen, Bavaria, Germany